CLINICAL TRIAL: NCT00612612
Title: A Phase 1 Study of Obatoclax Mesylate (GX15-070MS) in Combination With Fludarabine-Based Chemoimmunotherapy in Previously Treated Patients With B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Obatoclax, Fludarabine, and Rituximab in Treating Patients With Previously Treated Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00254; NCI-2009-00254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000582311; 07-100; 07-100 (Other: Dana-Farber Cancer Institute); 7945 (Other: CTEP); U01CA062490 (NIH); NCT00574938 (obsolete NCT alias)
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Leukemia; Prolymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, Prolymphocytic | interventions — obatoclax; fludarabine phosphate; Rituximab

ARMS (1):
- Treatment (obatoclax mesylate, fludarabine, rituximab) (Experimental): Patients receive obatoclax mesylate IV over 3 hours on days 1 and 3, fludarabine IV over 20-30 minutes on days 1-5, and rituximab IV over 4 hours on day 1 (days 1 and 3 of course 1 only). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients undergo peripheral blood collection for correlative studies. Samples are analyzed for expression of pro- and anti-apoptotic Bcl-2 family members by western blot; apoptosis induction by measurement of lymphocyte count, Annexin V staining, and Caspase and PARP cleavage; activated Bax by immunoprecipitation; and Bax promoter polymorphism by PCR amplification and direct sequencing.
  Interventions: Drug: obatoclax mesylate; Drug: fludarabine phosphate; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
Obatoclax may stop the growth of chronic lymphocytic leukemia by blocking blood flow to the cancer and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving obatoclax together with fludarabine and rituximab may kill more cancer cells. This phase I trial is studying the side effects and best dose of obatoclax when given together with fludarabine and rituximab in treating patients with B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose of obatoclax mesylate in combination with fludarabine phosphate-rituximab (FR) in patients with relapsed chronic lymphocytic leukemia.

SECONDARY OBJECTIVES:

I. To evaluate toxicity of obatoclax mesylate in combination with FR in this patient population.

II. To determine objective response rate and progression-free survival of obatoclax mesylate in combination with FR.

III. To correlate levels of anti-apoptotic Bcl-2 family members with drug response.

IV. To determine whether apoptosis is induced via the mitochondrial pathway in response to obatoclax mesylate and further enhanced by FR.

OUTLINE: This is a dose-escalation study of obatoclax mesylate.

Patients receive obatoclax mesylate IV over 3 hours on days 1 and 3, fludarabine IV over 20-30 minutes on days 1-5, and rituximab IV over 4 hours on day 1 (days 1 and 3 of course 1 only). Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo peripheral blood collection for correlative studies. Samples are analyzed for expression of pro- and anti-apoptotic Bcl-2 family members by western blot; apoptosis induction by measurement of lymphocyte count, Annexin V staining, and Caspase and PARP cleavage; activated Bax by immunoprecipitation; and Bax promoter polymorphism by PCR amplification and direct sequencing.

After completion of study therapy, patients are followed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of B-cell chronic lymphocytic leukemia (B-CLL) or prolymphocytic leukemia (PLL) arising from CLL
* No de novo PLL
* Malignant B cells must co-express CD5 with CD19 or CD20
* Patients who lack CD23 expression on their leukemia cells may not have t(11;14) or cyclin D1 overexpression, to rule out mantle cell lymphoma
* Must have documented lymphocytosis of > 5,000/uL
* Must require therapy based on any of the following criteria:

  * Massive or progressive splenomegaly and/or lymphadenopathy
  * Anemia (hemoglobin < 11 g/dL) or thrombocytopenia (platelet count < 100,000/uL)
  * Presence of weight loss > 10% over the preceding 6-month period
  * NCI grade 2 or 3 fatigue
  * Fevers > 100.5 F or night sweats for > 2 weeks without evidence of infection
* Progressive lymphocytosis with an increase of > 50% over a 2-month period or an anticipated doubling time of less than 6 months
* Must have received at least one prior therapy for B-CLL
* No known brain metastases
* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* Total bilirubin normal (unless due to Gilbert syndrome or compensated hemolysis)
* Life expectancy > 3 months
* Creatinine normal
* Fertile patients must use effective contraception
* Not pregnant or nursing
* Negative pregnancy test
* Any number of prior therapies allowed
* At least 1 year since prior fludarabine phosphate-rituximab combination therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No chemotherapy or radiotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* No other concurrent investigational agents
* AST and ALT < 2.5 times upper limit of normal
* Recovered from all prior therapy

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to obatoclax mesylate or other agents used in study
* Active Coombs' positive autoimmune hemolytic anemia
* Chronic active hepatitis B patients if not on appropriate antiviral therapy (e.g., lamivudine, adefovir)
* Other neurological disorders or dysfunction or a history of seizure disorder
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia including QTc > 450 msec
  * Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of obatoclax mesylate | 28 days
  DLT will be defined as any non-hematologic toxicity of grade 3 or greater severity (excluding asymptomatic grade 3 laboratory abnormalities that are not life-threatening and respond to treatment; grade 3 fatigue; grade 3 nausea, vomiting or diarrhea occurring without optimal prophylaxis; or expected grade 3 rituximab infusion reactions). Any grade 4 non-hematological toxicity, as well as any irreversible grade 2 cardiac, renal or neurologic toxicities, will be considered dose-limiting. Grading of non-hematologic toxicities will be according to NCI CTC version 3.0.

SECONDARY OUTCOMES:
Response evaluated using the Revised National Cancer Institute-sponsored Working Group Guidelines | Up to 2 years
  Described using descriptive statistics. Ninety-five percent confidence intervals will be calculated where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States